CLINICAL TRIAL: NCT06746688
Title: A First-In-Human Phase I, Open-Label, Dose-Escalating Trial to Assess the Safety, Tolerability and Immunogenicity/Preliminary Antitumor Activity of ES2B-C001 With or Without [Adjuvant] in HER2 Expressing Metastatic Breast Cancer
Brief Title: A First-in-human, Clinical Trial Assessing the Safety of ES2B-C001-S01 With or Without [Adjuvant] in Patients With HER2 Expressing Metastatic Breast Cancer.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ExpreS2ion Biotechnologies (Industry)
Collaborators: Gouya Insights (Unknown); VelaLabs (Unknown); KKS MedUni Vienna (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ES2B-C001-S01; 2024-516333-12-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-12; First posted 2024-12-24 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Breast Cancer Metastatic
Keywords: breast cancer; MBC; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: open-label, dose-escalating
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort C1: 50µg ES2B-C001 with [adjuvant] (Experimental)
  Interventions: Biological: ES2B-C001; Other: ISA 51 VD
- Cohort C2: 150µg ES2B-C001 with [adjuvant] (Experimental)
  Interventions: Biological: ES2B-C001; Other: ISA 51 VD
- Cohort C3: 450µg ES2B-C001 with [adjuvant] (Experimental)
  Interventions: Biological: ES2B-C001; Other: ISA 51 VD

INTERVENTIONS:
Biological: ES2B-C001 — Vaccine; Administration with or without [adjuvant] every third week for a total of five vaccinations.
Other: ISA 51 VD — Adjuvant; Administration together with ES2B-C001 every third week for a total of five vaccinations.

SUMMARY:
The trial is a first-in-human, phase I, open-label, dose-escalating trial to assess the safety and tolerability of ES2B-C001 combined with or without [adjuvant], in patients with human epidermal growth factor receptor 2 (HER2) expressing metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years at screening visit.
* Diagnosis of HER2-positive metastatic or locally advanced inoperable breast cancer (MBC).
* Life expectancy of at least 3 months.
* ECOG performance status 0-2.
* Patients have adequate bone marrow, kidney, liver, heart, and lung function without clinically significant laboratory parameters as judged by the investigator.
* 12-lead ECG without clinically significant abnormalities and no LBBB, QRS duration >140ms, or evidence of prior infarction.
* Recovered from side effects, adverse reactions, or adverse events due to prior therapy and/or surgery; any residual toxicities and toxicities related to current anticancer treatment must be ≤ Grade 2, except for alopecia, neuropathy or lymphoedema.
* If female, non-pregnant, postmenopausal, or practicing reliable contraception.
* If male, sterilized or using reliable contraception.

Exclusion Criteria:

* Any planned intravenous chemotherapy regimens or check point inhibitors, or previous therapy with those agents during the past 1 month and the patients are not neutropenic. For MBC maintenance therapy with a stable dose of HER2-directed mAbs or treatment with antibody drug conjugates (ADCs) at the discretion of the treating physician is allowed.
* Symptomatic CNS metastatic disease requiring treatment with high dose steroids (i.e., above 10 mg of prednisone or equivalent) within 14 days prior to first administration of ES2B-C001 (with or without adjuvant).
* Concurrent or recent (within 21 days or 5 half-lives) involvement in any other clinical trial with an investigational drug, device, or other experimental intervention.
* Concomitant severe or uncontrolled underlying medical and/or mental disease unrelated to the tumor, which in the opinion of the investigator is likely to compromise patient safety and affect the trial's outcome.
* Previous documented coronary artery disease or congestive heart failure (>NYHA II).
* Echocardiography with LVEF <55%.
* Uncontrolled hypertension.
* Active, known, or suspected autoimmune disease, except thyroid conditions sufficiently controlled on thyroid hormone therapy, and controlled insulin dependent diabetes.
* Necessity for long-term immunosuppression (≤ 4 mg dexamethasone may be used transiently).
* Systemic infection requiring intravenous antibiotics within 14 days before dosing.
* Chronic use of anti-viral agents, except for human immunodeficiency virus (HIV) or hepatitis B or C virus (HBV, HCV) treatments.
* History of severe hypersensitivity reactions to any of the trial drug components.
* Has received a live or live-attenuated vaccine within 30 days prior to the first dose of trial treatment. Note: Administration of inactivated or recombinant vaccines/killed vaccines are allowed.
* Birthmarks, tattoos, wounds, or skin conditions on deltoid region/buttocks that may obscure the assessment of injection site reactions.
* Female patients who are pregnant, or lactating.
* Any infection (including SARS-CoV-2), that in the opinion of the investigator would, upon inclusion in the trial, lead to potentially harming patients' safety or integrity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To determine the safety, tolerability, maximum tolerated dose (MTD) for ES2B-C001 alone or in combination with [adjuvant]. | From enrolment to the end of study at week 18
  * Nature and frequency of dose-limiting toxicities (DLTs).
  * Incidence, nature and severity of AEs graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
  * Incidence, nature and severity of injection site reactions according to FDA Guidance on Toxicity Grading Scales in Vaccine Trials (FDA, 2007).

SECONDARY OUTCOMES:
To investigate the immunogenicity of ES2B-C001 alone or in combination with [adjuvant]. | From enrolment to the end of study at week 18
  Immunogenicity as humoral immune response: Total anti-HER2 Immunoglobulin G (IgG) and IgG lambda titers in sera by enzyme-linked immunosorbent assay (ELISA).
To investigate the immunogenicity of ES2B-C001 alone or in combination with [adjuvant]. | From enrolment to the end of study at week 18
  Immunogenicity as humoral immune response: Optional: Isotyping of anti-HER2 Immunoglobulins in selected sera (e.g. IgM, IgG (IgG1-4), IgD, IgE, IgA).

OTHER OUTCOMES:
To determine the preliminary antitumor activity of ES2B-C001 alone or in combination with [adjuvant] observed. | From enrolment to the end of study at week 18
  Percentage of patients with measurable disease at baseline achieving Complete Remission (CR) or Partial Response (PR) according to RECIST 1.1 as assessed by the investigator during routine follow up.
To determine the preliminary antitumor activity of ES2B-C001 alone or in combination with [adjuvant] observed. | From enrolment to the end of study at week 18
  Percentage of patients with Disease Control Rate (DCR) according to RECIST 1.1 as assessed by the investigator during routine follow up.
To determine the preliminary antitumor activity of ES2B-C001 alone or in combination with [adjuvant] observed. | From enrolment to the end of study at week 18
  Progression free survival (PFS) in patients with Stable Disease (SD), or PR, at the time of first dosing of ES2B-C001 alone or in combination with [adjuvant] according to RECIST 1.1.
To determine the preliminary antitumor activity of ES2B-C001 alone or in combination with [adjuvant] observed. | From enrolment to the end of study at week 18
  Disease-free survival (DFS) in patients with CR at the time of first dosing of ES2B-C001 alone or in combination with [adjuvant] according to RECIST 1.1.
To determine the preliminary antitumor activity of ES2B-C001 alone or in combination with [adjuvant] observed. | From enrolment to the end of study at week 18
  Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas K. Jorgensen, Study Director — ExpreS2ion Biotechnologies
Locations (1):
- Medical University Of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Within the study de-identified patient data will be shared with
  * the operational study team, sponsor, auditor and for reporting of safety events to the regulatory agencies and EC
  * Data Monitoring Committees/ or other independent committees during the study
  * At the end - data listings are part of the Appendices of the CSR which will be shared to regulatory agencies and EC
Supporting Information: SAP, CSR